CLINICAL TRIAL: NCT02234791
Title: Mutation of the BTK Gene and Genotype-phenotype Correlation of Chinese Patients With X-Linked Agammaglobulinemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Principal Investigator, Chen Tongxin, Director of Allergy and Immunology department, Shanghai Children's Medical Center, Shanghai Children's Medical Center
Other Study IDs: BTK-20140828
Record Dates: First submitted 2014-08-29; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Agammaglobulinemia, BTK
MeSH Terms: conditions — Bruton type agammaglobulinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

GROUPS / COHORTS (1):
- gene mutation

SUMMARY:
X-linked agammaglobulinemia (XLA) is a humoral primary immunodeficiency in which affected patients have very low levels of peripheral B cells and a profound deficiency of all immunoglobulin isotypes. Mutations in the gene encoding for Bruton's tyrosine kinase (Btk) are responsible for most of the gammaglobulinemia.

We tend to investigate the gene mutation and clinical features of Chinese X-linked agammaglobulinemia (XLA) patients, and also examined the relationship between specific Btk gene mutations and severity of clinical presentation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of XLA A.male patients with less than 2% CD19-positive B cells; B.recurrent bacterial infection; C.decreased or absent immunoglobulins in serum

Exclusion Criteria for all groups:

* Presence of other primary immunodeficiency syndromes that do not meet the clinical and laboratory criteria for XLA

Ages: 1 Month to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: XLA patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
times of pneumonia | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children'S Medical Center, Shanghai, Shanghai Municipality, China